CLINICAL TRIAL: NCT03950466
Title: OBSTRUCTIVE SLEEP APNEA SYNDROME IN CHILDREN: HEALTH AND NEUROCOGNITIVE IMPACT. Real Life Pediatric Obstructive Sleep Apnea
Brief Title: Real Life Pediatric Obstructive Sleep Apnea
Acronym: RELIPOSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, ML Alonso-Alvarez, Principal Investigator, Medical Doctor, Sociedad Española de Neumología y Cirugía Torácica
Other Study IDs: PI 084-2016; STGRA17049OSASPAEDS-SH (Other Grant/Funding Number: Philips)
Record Dates: First submitted 2018-02-18; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Sleep Apnea, Obstructive; Children
Keywords: Sleep apnea; Children; Neurocognitive
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
OBJECTIVES:

PRIMARY: To analyze the cognitive alterations in children with Obstructive Sleep Apnea OSA in different age groups and changes at 12 months after treatment with a protocol based on usual clinical practice.

DESIGN:

Observational, longitudinal, prospective, and multicenter study.

DETAILED DESCRIPTION:
STUDY POPULATION: Children aged 3 to 12 years consecutively referred to the Sleep Units due to clinical suspicion of OSA.

SAMPLE SIZE: To evaluate the relationship between cognitive measures and polysomnographic variables and differences before-after treatment, a sample size of 1200 children is calculated.

METHODOLOGY: The followiong will be obtained in all children included in the study: personal medical history, Spanish version of Pediatric Sleep Questionnaire (PSQ), physical and otorhinolaryngological examination, neurocognitive assessment by customary neurocognitive and behavioral tests routinely used in Spain (CUMANIN neuropsychological tests, ENFEN neuropsychological tests, and Spanish version of the ECBI (Eyberg Child Behavior Inventory)), sleep study by polysomnography (PSG) or Respiratory Polygraphy (PR) and blood test.

The diagnosis and treatment of OSAS will be established according to the criteria of the Spanish Consensus Document of OSAS in children.

Depending on the treatment, three groups will be obtained: Group 1: Children with OSAS and adenotonsillar hypertrophy we will perform surgical treatment. Group 2: Children with OSAS and without adenotonsillar hypertrophy will be evaluated other treatments (sleep hygiene-diet and physical activity guidance, medical, orthodontic, continuous positive pressure on the airway (CPAP) treatment, Group 3: regular follow up but no treatment for children referred for suspicion of OSAS and that in PSG or RP the diagnosis of OSAS is not established. In all three groups, at 12 months, we will repeat all assessments as delineated for the initial visit

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 12 years consecutively referred to the Sleep Units due to clinical suspicion of OSA.

Exclusion Criteria:

* A significant medical and/or psychiatric comorbidity that may require urgent treatment (Respiratory Failure, Heart Failure, Cardiac Malformations, tumors, psychiatric type disorders that may require specific treatment…)
* Craniofacial malformations, deposit diseases and/or malformation syndromes (including Down's syndrome)
* Already diagnosed neurocognitive type disorders (e.g.: Autism, cerebral palsy, etc.)
* Attention deficit hyperactivity disorders previously diagnosed according to DSM-IV criteria
* Girls ≤ 12 with menarche at the time of starting the study
* Children that refuse to take part in the study (do not sign the Informed Consent

Ages: 3 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Children from 3 to 12 years-old referred consecutively to the Sleep Units of the participating sites due to clinical suspicion of OSA.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive changes after treatment in children with Obstructive Sleep Apnea (OSA) | 2018-2021
  Changes from before treatment in neurocognitive score on CUMANIN neuropsychological tests in chilren under 6 years old or ENFEN neuropsychological tests in children over six years old at 1 year after treatment

SECONDARY OUTCOMES:
Behavior changes after treatment in children with Obstructive Sleep Apnea (OSA) | 2018-2021
  Changes from before treatment in behavior score on ECBI (Eyberg Child Behavior Inventory) at 1 year after treatment
Sleep changes after treatment in children with Obstructive Sleep Apnea(OSA) | 2018-2021
  Changes from baseline in sleep study on polysomnography after treatment

CONTACTS AND LOCATIONS:
Overall Officials: María Luz Alonso-Alvarez, MD, Principal Investigator — Complejo Asistencial Universitario de Burgos
Locations (2):
- Spain (2):
  - Complejo Asistencial Universitario de Burgos, Burgos
  - Hospital Universitario de Burgos, Burgos